CLINICAL TRIAL: NCT00295152
Title: Effects of Community Occupational Therapy on the Daily Performance of Older Patients With Mild to Moderate Dementia and on the Sense of Competence of Their Primary Caregivers.
Brief Title: Effects of Community Occupational Therapy in Older Patients With Dementia and Their Caregivers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Alzheimer's Association (Other); VCVGZ Fund; (Unknown); Dutch Occupational Therapy Association (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: EDO project; Grant V-1999-023.
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2006-02

CONDITIONS: Community Occupational Therapy; Dementia Patients; Primary Caregivers of Dementia Patients
Keywords: elderly/aged; occupational therapy; daily activities; caregivers; sense of competence

INTERVENTIONS:
Behavioral: community occupational therapy in dementia

SUMMARY:
The purpose of this study is to determine the effects of community occupational therapy in older patients with mild ot moderate dementia and their primary caregivers.

DETAILED DESCRIPTION:
1. Objective To determine the effects of community occupational therapy on the daily performance of older patients with mild to moderate dementia and the sense of competence of their primary caregivers.
2. Methods

   1. design: a randomized controlled single-blind design is used with 3 measurement moments. We measure at baseline (before start of OT intervention), after 6 weeks (the effect measurement)and after 3 months after baseline (follow-up measurement).
   2. patients: 135 patients and their primary caregivers are needed to determine effects on the primary outcome measures of this intervention, with a power of 80% and alpha = 0.05/3. This power calculation is based on the outcomes of a pilot study (Graff, et al., 2003).
   3. intervention: 5 weeks client-centered community occupational therapy directed at both patients and primary caregivers using an OT guideline.The control group receives no OT intervention, but usual care.
   4. main outcome measures are: Assessment of Motor and Process Skills, Interview in Deterioration of Daily Activities in Dementia (IDDD)and Sense of Competence Questionnaire (SCQ)
   5. Analysis: analyses of covariance on intention-to-treat basis (Last Observation Carried Forward (LCOF))will be used to determine the effects of community OT on the daily performance of older patients with dementia and the sense of competence of their primary caregivers. Also secondary patients'and caregivers' health outcomes will be analyzed by analyses of covariance on intention-to-treat basis.
   6. Cost-effectiveness: the costs of this OT intervention will also be determined and a cost-effectiveness analysis will be carried out.

      3)Results: Results at baseline, at 6 weeks and at 3 months follow-up on primary outcome measures and on patients' and caregivers' secondary health outcomes and also the cost effectiveness of this intervention, will be analyzed and described in international publications.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* mild to moderate dementia (MMSE 10-24)
* living in the community at maximum of 50 kilometers from the Memory Clinic
* having an informal primary caregiver who was involved in the care for the patient at least once a week

Exclusion Criteria:

* depression: score > 12 on the Geriatric Depression Scale
* severe behavioral or psychological symptoms in dementia (BPSD) judged by a geriatrician
* severe illnesses, judged by a geriatrician
* no OT goals, determined by the researcher or research assistant
* caregivers having severe illnesses

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135
Dates: Start 2001-04; Study Completion 2005-02

PRIMARY OUTCOMES:
1.process skills scores of the patients on the Assessment of Motor and Process Skills (AMPS);
2. performance scores in daily activities of the patients on the Interview of Deterioration in Daily Activities in Dementia (IDDD);
3. Sense of competence scores of the primary caregivers on the Sense of Competence Questionnaire (SCQ).

SECONDARY OUTCOMES:
Patients:
1. motor skills scores on the AMPS
2. initiative in performing daily activities on the IDDD
3. general health scores on the General Health Questionnaire (GHQ-12)
4.Quality of life scored on the Dementia Quality of Life Instrument (DQOL)
5. Self-perception scores in occupational performance and satisfaction scores with this performance, scored on the Canadian Occupational Performance Measurement (COPM)
6. Mood/depression scored on the Cornell Depression Scale (CDS)
Caregiver:
1. mastery skills scored on the Mastery Scale
2. general health scores on the GHQ-12
3. quality of life scores on the DQOL
4. self-perception scores in occupational performance and satisfaction scores on the COPM
5. mood/depression scores on the Center for Epidemiologic Studies Depression Scales (Ces-D)
6. Copings skills scores on the JCS

CONTACTS AND LOCATIONS:
Overall Officials: Marcel GM Olde-Rikkert, PhD, MD, Principal Investigator — Department of Geriatrics Radboud University Nijmegen Medical Centre
Locations (1):
- Memory Clinic and Geriatic Department Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Gitlin LN, Winter L, Corcoran M, Dennis MP, Schinfeld S, Hauck WW. Effects of the home environmental skill-building program on the caregiver-care recipient dyad: 6-month outcomes from the Philadelphia REACH Initiative. Gerontologist. 2003 Aug;43(4):532-46. doi: 10.1093/geront/43.4.532. PMID 12937332
- [Background] Steultjens EM, Dekker J, Bouter LM, Jellema S, Bakker EB, van den Ende CH. Occupational therapy for community dwelling elderly people: a systematic review. Age Ageing. 2004 Sep;33(5):453-60. doi: 10.1093/ageing/afh174. PMID 15315918
- [Background] Vernooij-Dassen MJ, Felling AJ, Brummelkamp E, Dauzenberg MG, van den Bos GA, Grol R. Assessment of caregiver's competence in dealing with the burden of caregiving for a dementia patient: a Short Sense of Competence Questionnaire (SSCQ) suitable for clinical practice. J Am Geriatr Soc. 1999 Feb;47(2):256-7. doi: 10.1111/j.1532-5415.1999.tb04588.x. No abstract available. PMID 9988301
- [Background] Vernooij-Dassen M, Lamers C, Bor J, Felling A, Grol R. Prognostic factors of effectiveness of a support program for caregivers of dementia patients. Int J Aging Hum Dev. 2000;51(4):259-74. doi: 10.2190/P8L1-N8QD-VTJ4-EURT. PMID 11246648
- [Background] Teunisse S, Derix MM. The interview for deterioration in daily living activities in dementia: agreement between primary and secondary caregivers. Int Psychogeriatr. 1997;9 Suppl 1:155-62. doi: 10.1017/s1041610297004845. PMID 9447438
- [Result] Graff MJL, et al.Occupational therapy at home for older individuals with mild to moderate cognitive impairments and their primary caregivers: a pilot study. Occupational Therapy Journal of Research 23, 155-163, 2003.
- [Result] Graff MJL, Melick van MBM. The development, testing and implementation of an occupational therapy guideline. The guideline for the OT diagnosis and treatment of older persons with cognitive impairments. Ducth Occupational Therapy Journal 28, 169-174, 2000.
- [Result] Melick van MBM, Graff MJL. Occupational therapy for geriatric patients. The guideline for occupational therapy in geriatric patients with mild to moderate cognitive impairments. Dutch Journal of Occupational Therapy 28, 176-181, 2000
- [Result] Graff MJL, et al. How can occupational therapy improve the daily performance and communication of an older patient with dementia and his primary caregiver: a case study. Dementia: the journal of social research and practice. 2006. In press.
- [Derived] Graff MJ, Vernooij-Dassen MJ, Thijssen M, Dekker J, Hoefnagels WH, Rikkert MG. Community based occupational therapy for patients with dementia and their care givers: randomised controlled trial. BMJ. 2006 Dec 9;333(7580):1196. doi: 10.1136/bmj.39001.688843.BE. Epub 2006 Nov 17. PMID 17114212